CLINICAL TRIAL: NCT05940623
Title: Impact of Home Intraocular Pressure Telemonitoring on Intraocular Pressure Control and Glaucoma Progression - A Randomized Control Trial
Brief Title: Impact of Home Intraocular Pressure Telemonitoring on Intraocular Pressure Control and Glaucoma Progression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Icare Finland Oy (Industry)
Responsible Party: Principal Investigator, Professor Christopher K.S. Leung, Clinical Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Protocol_iCare_v2_20230523
Record Dates: First submitted 2023-07-04; First posted 2023-07-11 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Glaucoma; Intraocular Pressure; Primary Open Angle Glaucoma
Keywords: Ophthalmology; Glaucoma
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle

STUDY DESIGN:
Intervention Model Description: iCare Home2 tonometer
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Management Paradigm I: Standard care and home IOP telemonitoring with smart phone-based intervention (Active Comparator): Eligible patients randomized to Management Paradigm I will be provided with an iCare Home and instructed to measure and upload 6 IOP measurements weekly (2 days a week, 1 measurement in the early morning (5 am to 9 am), 1 during the mid-day (12 pm to 4 pm) and 1 in the evening (7 pm to 11pm)) to a secure server via iCare. Patients will be treated with topical prostaglandin analogue after baseline IOP measurements. A text message will be sent to the patient's smart phone to (1) inform whether the treatment goal is achieved over the past 4 weeks (i.e., ≥75% of the self- measured IOP measurements are below the target IOP) and (2) remind adherence to medications. The patients will need to reply via a text message reporting how many times eyedrops are missed over the past 4 weeks. A nurse will phone the patient if a reply message is not received or the number of home IOP measurements is less than 20 over the past 4 weeks.
  Interventions: Device: Standard care and home IOP telemonitoring with smart phone-based intervention
- Management paradigm II: Standard care and smart phone-based intervention (No Intervention): Patients will be treated with a topical prostaglandin analogue after baseline IOP measurements (described below). Additional treatment will be provided in the following order: carbonic anhydrase inhibitor, brimonidine, beta blocker, and selective laser trabeculoplasty (SLT) when the target IOP is not achieved. Fixed combination will be given whenever possible to improve adherence. Similar to Management Paradigm I, smart phone-based intervention includes (1) a text message from the investigators to inform whether the target pressure is attained (with reference to the latest clinic GAT measurement) and remind medication adherence every 4 weeks and (2) a reply message from the patients regarding how many times eyedrops are missed over the past 4 weeks.

INTERVENTIONS:
Device: Standard care and home IOP telemonitoring with smart phone-based intervention — We expect that (1) GAT measurements over 30 months of follow-up for patients randomized to Management Paradigm I to be smaller compared with those randomized to Management Paradigm II; and that (2) the rates of RNFL/GCIPL thinning would be slower for those randomized to Management Paradigm I compared with those randomized to Management Paradigm II
  Arms: Management Paradigm I: Standard care and home IOP telemonitoring with smart phone-based intervention

SUMMARY:
The goal of this clinical trial is to conduct a study randomizing glaucoma patients to home intra-ocular pressure (IOP) telemonitoring combined with Smart phone-based intervention (Management Paradigm I) or Smart phone-based intervention alone (Management Paradigm II), with the objectives to compare (1) Goldmann applanation tonometry (GAT) intra-ocular pressure (IOP) measurements over the entire study period (primary outcome measure) and (2) the rates of Retinal nerve fiber layer (RNFL) thinning (secondary outcome measure) between the two Management Paradigms. We hypothesize that glaucoma patients randomized to Management Paradigm I will (1) attain lower levels of intra-ocular pressure (IOP), and (2) a slower rate of Retinal nerve fiber layer (RNFL) and ganglion cell inner plexiform layer (GCIPL) thinning compared with those randomized to Management Paradigm II because of having a more precise assessment of intra-ocular pressure (IOP) to guide intra-ocular pressure (IOP)- lowering therapy would be feasible in Management Paradigm I.

It aims to:

to compare (1) Goldmann applanation tonometry (GAT) intra-ocular pressure (IOP) measurements over the entire study period (primary outcome measure) and (2) the rates of Retinal Nerve Fiber Layer (RNFL) thinning (secondary outcome measure) between the two Management Paradigms.

Participants will asked to do,

* Management Paradigm I: will be provided with an iCare Home and instructed to measure and upload 6 intra-ocular pressure (IOP) measurements weekly (2 days a week, 1 measurement in the early morning (5 am to 9 am), 1 during the mid-day (12 pm to 4 pm) and 1 in the evening (7 pm to 11pm)) to a secure server via iCare CLINIC (the number of weekly intra-ocular pressure (IOP) measurements follows the number of weekly blood pressure measurements in the HyperLink study). The morning measurement will include two readings with the first obtained in the supine position before getting out of the bed and the second obtained in the upright position right after. Patients may take additional intra-ocular pressure (IOP) measurements in supine position if they wake up in bed from sleep, as well as other times of the day, but this is not mandatory. These additional intra-ocular pressure (IOP) measurements will not be included for treatment decisions during the study period.
* Management paradigm II: Patients will be treated with a topical prostaglandin analogue after baseline intra-ocular pressure (IOP) measurements.

DETAILED DESCRIPTION:
Study design This is a 30-month prospective, multicenter, randomized clinical trial to compare the treatment outcomes between two management paradigms: (I) home IOP telemonitoring combined with smart phone-based intervention, and (II) standard care plus smart phone- based intervention, in 142 patients with newly diagnosed primary open-angle glaucoma (POAG). Both management paradigms aim to decrease the IOP by the same degree according to the disease severity. For mild to moderate glaucoma (visual field MD ≥ -12 dB), we aim to decrease the IOP by at least 20% from the baseline (methods of baseline IOP measurements are described below) targeting the IOP levels <21 mmHg; for advanced glaucoma (visual field MD <-12 dB), we aim to decease the IOP by at least 25% from the baseline targeting the IOP levels <15 millimeters of mercury (mmHg). The unit of observation for sample size estimation and randomization will be based on subject. Patients will be randomized by minimization, stratified by demographics (age, gender, and axial length) and clinical parameters (baseline IOP levels and baseline RNFL thickness of the better eye). For analysis of outcome measures, both eyes will be included if both eyes are eligible for inclusion (described below), taking account for clustering between fellow eyes. Intent-to-treat analyses will be performed. The primary outcome measure will be clinic-measured GAT measurements collected at 3-month intervals over 30 months of study follow-up. The secondary outcome measures include the rates of change of global, superotemporal and inferotemporal RNFL thicknesses, and the rates of change of global and regional GCIPL thicknesses. We expect that (1) GAT measurements over 30 months of follow-up for patients randomized to Management Paradigm I to be smaller compared with those randomized to Management Paradigm II; and that (2) the rates of RNFL/GCIPL thinning would be slower for those randomized to Management Paradigm I compared with those randomized to Management Paradigm II. Additional analyses include (i) comparisons of visual field (VF) survival probabilities (defined by the Early Manifest Glaucoma Trial (EMGT) criteria) and (ii) the number of ocular hypotensive medications between the treatment groups during the study follow-up; and (iii) investigation of risk factors associated with the rate of RNFL/GCIPL thinning including mean IOP (measured by iCare Home or GAT), long-term IOP fluctuations (IOP deviated from the mean during study follow-up), and glaucoma severity (baseline average RNFL thickness). Study safety endpoints will include: (i) visual field (VF) progression; (ii) decrease in visual acuity (VA) ≥2 lines; and (iii) IOP≥35mmHg on 2 consecutive visits. Patients will exit the study and receive additional treatment(s) if any of the study safety endpoints is reached. Patients randomized to have IOP measured by iCare Home will continue the home IOP measurements until the completion of study. All patients in Management Paradigms I and II will be followed up 3-monthly in the clinic for GAT, optical coherence tomography retinal nerve fiber layer (OCT RNFL) imaging and perimetry.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed primary open-angle glaucoma (POAG)
* Best corrected visual acuity (VA) ≥20/40 for the included eye(s)

Exclusion Criteria:

* IOP >35 millimeters of mercury (mmHg)
* Dry eye syndrome
* Central corneal thickness <500μm or >600μm
* Failure to complete the iCare Home certification procedure at the baseline visits
* Only one eye with functional vision
* Inability to perform reliable visual field (VF)
* Pathological myopia (eyes with axial length≥26mm with lacquer cracks and chorioretinal atrophy)
* Suboptimal quality of optical coherence tomography (OCT) images (described below in RNFL imaging)
* Previous intraocular surgery or corneal refractive surgery other than uncomplicated cataract extraction
* Diabetic retinopathy/maculopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2023-08-24 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinic-measured Goldmann applanation tonometry measurements collected at 3-month interval over 30 months of study follow-up. | From baseline to 30 months, at 3-month intervals
  Goldmann applanation tonometry is an instrument measures intra-ocular pressure based on Imbert-Fick law. The Goldmann equation states: Po = (F/C) + Pv [Po is the IOP in millimeters of mercury (mmHg), F is the rate of aqueous formation, C is the facility of outflow, and Pv is the episcleral venous pressure].

SECONDARY OUTCOMES:
Rate of changes of global, superotemporal and inferotemporal Retinal Nerve Fiber Layer (RNFL) thickness, and the rate of changes of global and regional Ganglion cell-inner plexiform layer (GCIPL) thickness. | From baseline to 30 months, at 3-month intervals
  RNFL and GCIPL thickness could be assessed by Optical coherence tomography (OCT), which analyze the temporal delay of backscattered light from tissue structures.
  RNFL thickness (µm) could be measured by an optic disc cube OCT scan. RNFL thickness is presented on 2 circular charts, 1 with 12 equal sized sectors, and the other with 4 equal sectors each representing 1 quadrant (superior, nasal, temporal and inferior).
  GCIPL thickness (µm) could be measured by a macular OCT scan. GCIPL thickness is presented on a thickness map, with 6 equal sized sectors.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Leung, Principal Investigator — The University of Hong Kong

IPD SHARING:
Plan to Share IPD: No
Our plan is focused on publishing the analyzed results of our research through peer-review, journals and conference papers. We understand the importance of patient privacy and confidentiality. Therefore, we will not share any individual patient data with any third parties.

REFERENCES:
- [Background] Flaxman SR, Bourne RRA, Resnikoff S, Ackland P, Braithwaite T, Cicinelli MV, Das A, Jonas JB, Keeffe J, Kempen JH, Leasher J, Limburg H, Naidoo K, Pesudovs K, Silvester A, Stevens GA, Tahhan N, Wong TY, Taylor HR; Vision Loss Expert Group of the Global Burden of Disease Study. Global causes of blindness and distance vision impairment 1990-2020: a systematic review and meta-analysis. Lancet Glob Health. 2017 Dec;5(12):e1221-e1234. doi: 10.1016/S2214-109X(17)30393-5. Epub 2017 Oct 11. PMID 29032195
- [Background] Quigley HA, Broman AT. The number of people with glaucoma worldwide in 2010 and 2020. Br J Ophthalmol. 2006 Mar;90(3):262-7. doi: 10.1136/bjo.2005.081224. PMID 16488940
- [Background] Weinreb RN, Leung CK, Crowston JG, Medeiros FA, Friedman DS, Wiggs JL, Martin KR. Primary open-angle glaucoma. Nat Rev Dis Primers. 2016 Sep 22;2:16067. doi: 10.1038/nrdp.2016.67. PMID 27654570
- [Background] Liu JH, Zhang X, Kripke DF, Weinreb RN. Twenty-four-hour intraocular pressure pattern associated with early glaucomatous changes. Invest Ophthalmol Vis Sci. 2003 Apr;44(4):1586-90. doi: 10.1167/iovs.02-0666. PMID 12657596
- [Background] Liu JH, Sit AJ, Weinreb RN. Variation of 24-hour intraocular pressure in healthy individuals: right eye versus left eye. Ophthalmology. 2005 Oct;112(10):1670-5. doi: 10.1016/j.ophtha.2005.05.007. PMID 16095707
- [Background] Liu JH, Kripke DF, Twa MD, Hoffman RE, Mansberger SL, Rex KM, Girkin CA, Weinreb RN. Twenty-four-hour pattern of intraocular pressure in the aging population. Invest Ophthalmol Vis Sci. 1999 Nov;40(12):2912-7. PMID 10549652
- [Background] Bengtsson B, Leske MC, Hyman L, Heijl A; Early Manifest Glaucoma Trial Group. Fluctuation of intraocular pressure and glaucoma progression in the early manifest glaucoma trial. Ophthalmology. 2007 Feb;114(2):205-9. doi: 10.1016/j.ophtha.2006.07.060. Epub 2006 Nov 13. PMID 17097736
- [Background] Caprioli J, Coleman AL. Intraocular pressure fluctuation a risk factor for visual field progression at low intraocular pressures in the advanced glaucoma intervention study. Ophthalmology. 2008 Jul;115(7):1123-1129.e3. doi: 10.1016/j.ophtha.2007.10.031. Epub 2008 Feb 20. PMID 18082889
- [Background] Barkana Y, Anis S, Liebmann J, Tello C, Ritch R. Clinical utility of intraocular pressure monitoring outside of normal office hours in patients with glaucoma. Arch Ophthalmol. 2006 Jun;124(6):793-7. doi: 10.1001/archopht.124.6.793. PMID 16769832
- [Background] Hughes E, Spry P, Diamond J. 24-hour monitoring of intraocular pressure in glaucoma management: a retrospective review. J Glaucoma. 2003 Jun;12(3):232-6. doi: 10.1097/00061198-200306000-00009. PMID 12782841
- [Background] Schwartz GF, Quigley HA. Adherence and persistence with glaucoma therapy. Surv Ophthalmol. 2008 Nov;53 Suppl1:S57-68. doi: 10.1016/j.survophthal.2008.08.002. PMID 19038625
- [Background] Leske MC, Heijl A, Hussein M, Bengtsson B, Hyman L, Komaroff E; Early Manifest Glaucoma Trial Group. Factors for glaucoma progression and the effect of treatment: the early manifest glaucoma trial. Arch Ophthalmol. 2003 Jan;121(1):48-56. doi: 10.1001/archopht.121.1.48. PMID 12523884
- [Background] Garway-Heath DF, Crabb DP, Bunce C, Lascaratos G, Amalfitano F, Anand N, Azuara-Blanco A, Bourne RR, Broadway DC, Cunliffe IA, Diamond JP, Fraser SG, Ho TA, Martin KR, McNaught AI, Negi A, Patel K, Russell RA, Shah A, Spry PG, Suzuki K, White ET, Wormald RP, Xing W, Zeyen TG. Latanoprost for open-angle glaucoma (UKGTS): a randomised, multicentre, placebo-controlled trial. Lancet. 2015 Apr 4;385(9975):1295-304. doi: 10.1016/S0140-6736(14)62111-5. Epub 2014 Dec 19. PMID 25533656
- [Background] Meier-Gibbons F, Berlin MS, Toteberg-Harms M. Twenty-four hour intraocular pressure measurements and home tonometry. Curr Opin Ophthalmol. 2018 Mar;29(2):111-115. doi: 10.1097/ICU.0000000000000460. PMID 29278546
- [Background] Xu SC, Gauthier AC, Liu J. The Application of a Contact Lens Sensor in Detecting 24-Hour Intraocular Pressure-Related Patterns. J Ophthalmol. 2016;2016:4727423. doi: 10.1155/2016/4727423. Epub 2016 Jul 25. PMID 27525110
- [Background] Mudie LI, LaBarre S, Varadaraj V, Karakus S, Onnela J, Munoz B, Friedman DS. The Icare HOME (TA022) Study: Performance of an Intraocular Pressure Measuring Device for Self-Tonometry by Glaucoma Patients. Ophthalmology. 2016 Aug;123(8):1675-1684. doi: 10.1016/j.ophtha.2016.04.044. Epub 2016 Jun 9. PMID 27289178
- [Background] Margolis KL, Asche SE, Bergdall AR, Dehmer SP, Groen SE, Kadrmas HM, Kerby TJ, Klotzle KJ, Maciosek MV, Michels RD, O'Connor PJ, Pritchard RA, Sekenski JL, Sperl-Hillen JM, Trower NK. Effect of home blood pressure telemonitoring and pharmacist management on blood pressure control: a cluster randomized clinical trial. JAMA. 2013 Jul 3;310(1):46-56. doi: 10.1001/jama.2013.6549. PMID 23821088
- [Background] Margolis KL, Asche SE, Dehmer SP, Bergdall AR, Green BB, Sperl-Hillen JM, Nyboer RA, Pawloski PA, Maciosek MV, Trower NK, O'Connor PJ. Long-term Outcomes of the Effects of Home Blood Pressure Telemonitoring and Pharmacist Management on Blood Pressure Among Adults With Uncontrolled Hypertension: Follow-up of a Cluster Randomized Clinical Trial. JAMA Netw Open. 2018 Sep 7;1(5):e181617. doi: 10.1001/jamanetworkopen.2018.1617. PMID 30646139
- [Background] Yu M, Lin C, Weinreb RN, Lai G, Chiu V, Leung CK. Risk of Visual Field Progression in Glaucoma Patients with Progressive Retinal Nerve Fiber Layer Thinning: A 5-Year Prospective Study. Ophthalmology. 2016 Jun;123(6):1201-10. doi: 10.1016/j.ophtha.2016.02.017. Epub 2016 Mar 19. PMID 27001534
- [Background] Lin C, Mak H, Yu M, Leung CK. Trend-Based Progression Analysis for Examination of the Topography of Rates of Retinal Nerve Fiber Layer Thinning in Glaucoma. JAMA Ophthalmol. 2017 Mar 1;135(3):189-195. doi: 10.1001/jamaophthalmol.2016.5111. PMID 28152147
- [Background] Bodenheimer T, Wagner EH, Grumbach K. Improving primary care for patients with chronic illness. JAMA. 2002 Oct 9;288(14):1775-9. doi: 10.1001/jama.288.14.1775. PMID 12365965
- [Background] Heijl A, Leske MC, Bengtsson B, Bengtsson B, Hussein M; Early Manifest Glaucoma Trial Group. Measuring visual field progression in the Early Manifest Glaucoma Trial. Acta Ophthalmol Scand. 2003 Jun;81(3):286-93. doi: 10.1034/j.1600-0420.2003.00070.x. PMID 12780410
- [Background] Tu XM, Kowalski J, Zhang J, Lynch KG, Crits-Christoph P. Power analyses for longitudinal trials and other clustered designs. Stat Med. 2004 Sep 30;23(18):2799-815. doi: 10.1002/sim.1869. PMID 15344187
- [Background] Nakakura S, Asaoka R, Terao E, Nagata Y, Fukuma Y, Oogi S, Shiraishi M, Kiuchi Y. Evaluation of rebound tonometer iCare IC200 as compared with IcarePRO and Goldmann applanation tonometer in patients with glaucoma. Eye Vis (Lond). 2021 Jul 1;8(1):25. doi: 10.1186/s40662-021-00249-z. PMID 34193284
- [Background] Badakere SV, Chary R, Choudhari NS, Rao HL, Garudadri C, Senthil S. Agreement of Intraocular Pressure Measurement of Icare ic200 with Goldmann Applanation Tonometer in Adult Eyes with Normal Cornea. Ophthalmol Glaucoma. 2021 May-Jun;4(3):238-243. doi: 10.1016/j.ogla.2021.04.002. PMID 34030826
- See also: 510(K) Summary of safety and effectiveness for iCare Home tonometer — https://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfpmn/pmn.cfm?ID=K163343.